CLINICAL TRIAL: NCT02522390
Title: The Nutrition Researcher Cohort 2014 Study; New Standardized Self-quantification Methodologies Serving Both Research and Personal Health Maintenance
Brief Title: The Nutrition Researcher Cohort 2014 Study
Acronym: NRC250
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: TNO (Other)
Collaborators: University of Eastern Finland (Other); Lund University (Other); NIHS (Unknown); University of Barcelona (Other); University College Dublin (Other); Newcastle University (Other); Technical University Munchen (Unknown); Universitaire Ziekenhuizen KU Leuven (Other); University of Oslo (Other); University of Copenhagen (Other); University of Graz (Other); Tufts University (Other); Charles University, Czech Republic (Other); NuGo (Unknown); VITAS Analytical Services (Unknown); Humboldt-Universität zu Berlin (Other); CSIRO Animal, Food and Health Sciences (Unknown); SwissAnalysis AG (Unknown); Agroscope Liebefeld-Posieux Research Station ALP (Other); CRA NUT - Centro di Ricerca per gli Alimenti e la Nutrizione (Unknown)
Responsible Party: Principal Investigator, Ivana Bobeldijk-Pastorova, Project Manager, TNO
Other Study IDs: P9616
Record Dates: First submitted 2015-03-23; First posted 2015-08-13 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Nutritional Physiological Phenomena; Health; Biological Markers
Keywords: data collection; personal health services; personal health records; do-it-yourself; nutrition researchers; cohort studies; databases, factual; self-quantification methods
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — "do-it-yourself", at-home measurements of blood glucose and blood cholesterol.
  In addition, the plasma metabolome and selected biomarkers (from dried blood spot), urinary metabolome (from collected urine), DNA damage (from dried blood spots, telomere length and mitochondrial DNA deletions, DNA base damage/oxidation, gamma H2AX DNA strand break assay), micronutrient analysis (from dried blood spot or capillary blood collection) and microbiome (sequencing metagenomics/Fecal Swabs) will be offered to participants as additional measurements, if funding or in-kind sponsoring is available.
  Funding is already available for:
  * Dried blood spot collection for analysis of biomarkers (including fatty acids, vitamins, amino acids) and metabolomics;
  * Faecal collection (swab) for metagenome analysis
  * Capillary blood collection for CRP, HbA1c and other parameters
  * OGTT sampling kit for analysis of insulin and c-peptide;
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nutrition Researcher Cohort: This cohort study is an observational, one-group study. The intervention consists of research activities that participants are asked to perform throughout the cohort, including the use of do-it-yourself devices, filling out online-questionnaires and sample collection with supplied kits for the analysis of various health parameters. The frequency with which participants are asked to measure these health parameters varies, ranging from once to weekly.
  Interventions: Other: Research activities

INTERVENTIONS:
Other: Research activities — Measurements are primarily based on "do-it-yourself" non-invasive or minimally invasive methods. Participants upload collected data to the Personal Health Portal.
  The measurements are divided into required and optional measurements. The required measurements mainly include routine methodology (e.g. weight, blood pressure, blood glucose); the latter also include methods under development that will be fine-tuned along the project. Which additional measures will be offered to participants is dependent on if funding or in-kind sponsoring is available. Participants will receive measurement kits for these analyses at-home and will be responsible for collection, labeling and shipment of samples themselves. After analysis the resulting data are uploaded to the user accounts.
  Other Names: Do-it-yourself devices; filling out online-questionnaires; sample collection with supplied kits

SUMMARY:
The primary objective of the planned Nutrition Research Cohort (NRC) n250 study is to develop and evaluate the open access Nutrition Researcher Cohort for gathering personal health data from nutrition researchers, including analytical methods, standards and operation procedures, data infrastructure, ethical and privacy aspects, and governance.

Besides, the study aims to exploit and analyse data on food, nutrient and bioactive compound intake and exposure, biomarkers for food, health and/or disease and health and/or disease related measurements to study the relation between nutrition, health and development of disease (on individual level).

In addition, data will be used to develop applications that visualise personal health risks based for example on (validated) recommendations and applications that predict individual health risks.

The study is designed as an open, one-group, exploratory cohort study. The total NRC cohort will be composed of about 250 life sciences employees and students from different, predominantly European, countries. This allows optimal involvement of participants in shaping all aspects of the cohort and the ownership of data. We aim to recruit about in total 20 male and female scientists per participating country.

DETAILED DESCRIPTION:
The NRC n250 study is an open, one-group, open-ended cohort study, which will include participants from 10 different countries. The study will be coordinated by national contact points from each of the participating countries.

The NRC cohort study will start early 2015 and continue developing from that moment on. Recruitment will start immediately after approval of the study protocol in the country where it has been submitted. The Participant Information Form, which contains the complete research protocol as developed by the consortium partners, is available online via the NRC website. This way, potential participants can make an informed decision on whether or not they want to participate.

The NRC n250 study will provide a dataset from 250 individuals, including food intake, microbiome composition, oral glucose tolerance tests, a series of plasma (bio)chemistry outcomes, plasma and urine metabolome and DNA damage, together with anthropometrics and life style questionnaires.

Since the aim is to build up a powerful open access cohort, there is no end-date defined for this study. The collected data will be used for various analyses on food intake, biomarkers for food intake and/or health and/or disease, and health/disease related measurements.

The research questions that will be answered with this cohort are largely not known yet, since it is not known which data will become available. A NRC Scientific committee is established to judge whether or not the data in the cohort may be used for answering the proposed research questions. This Scientific committee consists of the principal investigators of the individual participating countries.

The Scientific committee is the entity that views all proposals (new studies, research questions) and decides whether or not it is in line with aim of NRC as well as ethics as well as scientifically robust. Approval for proposals can be obtained by positive response from a majority of the members (quality and ethics of proposals).

Institutions/companies that obtain data for a specific proposal, are only allowed to use the data for that specific purpose.

The NRC cohort also aims to serve as a platform to validate specific questionnaires (including food intake) or additional measurements (that are within scope of the NRC objectives). For offering an additional measurement or questionnaire to participants for health parameters that are already included in the protocols, also a request for approval should be filed to the scientific committee. The scientific committee will then decide (based on a positive response of the majority of the committee) if this measurement or questionnaire may be added. A request for data analysis with these new measures or questionnaires, other than validation purposes, has to be filed separately. If a request for approval is granted, participants still have the opportunity to opt out their data for use for this purpose.

For research questions that require additional measurements for health parameters that are not yet included in the protocol, amendments will be submitted to the Dutch Medical Research and Ethics Committee (MREC).

ELIGIBILITY:
Inclusion Criteria:

* Employees or students that are active in the field of nutrition and/or biology and/or health (e.g. epidemiologists, dieticians, nutrition students and researchers) that have a basic knowledge of nutrition and/or human biology and are thus able to form a scientific judgement on his/her own health data;
* good understanding of the English written language, since all communication is handled in English.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The NRC cohort will be composed of employees and students in the area of life sciences. This allows optimal involvement of participants in shaping all aspects of the cohort and the ownership of data. We aim to recruit about 250 male and female scientists for the entire cohort. For each participating country it is aimed to recruit about 25 participants, taking drop-out and varying submission and/or starting dates between the 15 participating countries into account. Besides, a higher number of participants will increase the chance of being able to compare the data with other countries.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2015-01; Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Body height | Baseline (week 1)
  measured with do-it-yourself device in at-home setting
Body weight | Each week during entire cohort (five years in total)
  measured with do-it-yourself device in at-home setting
Single Nucleotide Polymorphism (SNP) profile | Once during the cohort at baseline (a timepoint chosen by the participant in the first three months of the cohort)
  No specific time of measurement has to be specified as genetic profile is not subject to change
Waist-to-hip ratio | Monthly during entire cohort (Month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 for each year of the five year cohort)
  measured with waist circumference and hip circumference; measured with centimeter in at-home setting
Blood pressure | Monthly during entire cohort (Month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 for each year of the five year cohort)
  Diastolic and systolic blood pressure; measured with do-it-yourself device in at-home setting
Resting heart rate | Monthly during entire cohort (Month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 for each year of the five year cohort)
  measured after sitting still for at least 5 minutes; measured with do-it-yourself device in at-home setting
fasting blood glucose | Monthly during entire cohort (Month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 for each year of the five year cohort)
  measured after 8h fasting (only drinking water is allowed); measured with do-it-yourself device in at-home setting
Blood cholesterol | quarterly during entire cohort (Month 3, M6, M9, M12 for each year of the five year cohort)
  HDL, LDL, total cholesterol, triglycerides; measured with do-it-yourself device in at-home setting
Food intake | quarterly during entire cohort (Month 3, M6, M9, M12 for each year of the five year cohort)
  registration of food intake during two weekdays and one weekend day via an online application (e.g. FatSecret)
Physical activity tracker | quarterly during entire cohort (Month 3, M6, M9, M12 for each year of the five year cohort)
  Registration of physical activity with a physical activity tracker (e.g. FitBit) for at least one week continuously

SECONDARY OUTCOMES:
biomarker profile | once, at baseline (at a timepoint chosen by the participant in the first three months of the cohort); this measure will be repeated only if funding for analysis becomes available
  biomarkers for food intake (vitamins, fatty acids) and other blood biomarkers (cortisol, C Reactive protein (CRP), thyroid stimulating hormone (TSH), etc.)
do-it-yourself oral glucose tolerance test | once, at baseline (at a timepoint chosen by the participant in the first three months of the cohort); this measure will be repeated only if funding for analysis becomes available
  insulin, glucose, c-peptide, HbA1c; including response profile after oral glucose tolerance test
metabolomics | once, at baseline (at a timepoint chosen by the participant in the first three months of the cohort); this measure will be repeated only if funding for analysis becomes available
metagenome | once, at baseline (at a timepoint chosen by the participant in the first three months of the cohort); this measure will be repeated only if funding for analysis becomes available
general health status | once per year during entire cohort (Month 12, M24, M36, M48, M60)
  via a questionnaire
lifestyle (smoking, alcohol consumption, etc.) | once per year during entire cohort (Month 12, M24, M36, M48, M60)
  via a questionnaire
general food intake | once per year during entire cohort (Month 12, M24, M36, M48, M60)
  via a food frequency questionnaire
quality of sleep | once per year during entire cohort (Month 12, M24, M36, M48, M60)
  via a questionnaire
stress questionnaire | once per year during entire cohort (Month 12, M24, M36, M48, M60)
physical activity | once per year during entire cohort (Month 12, M24, M36, M48, M60)
  via a questionnaire
wellness | once per year during entire cohort (Month 12, M24, M36, M48, M60)
  via a questionnaire
cognition | once per year during entire cohort (Month 12, M24, M36, M48, M60)
  via a questionnaire
quality of life | once per year during entire cohort (Month 12, M24, M36, M48, M60)
  via a questionnaire

OTHER OUTCOMES:
compliance with the study protocol | after one year (june 2016)
  compliance will be determined for each of the included measurements and compared between participating countries
user experiences with participating in the cohort | after one year (june 2016)
  as measured via a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: André Boorsma, PhD, Principal Investigator — TNO; Baukje de Roos, Principal Investigator — Newcastle University; Giuditta Perozzi, Principal Investigator — CRA-NUT; Lorraine Brennan, Principal Investigator — University College Dublin; Christophe Matthys, Principal Investigator — University Leuven; Irina Dobre, Principal Investigator — University of Copenhagen; Miroslav Petr, Principal Investigator — Charles University Prague; Andre Mazur, Principal Investigator — INRA - French National Institute for Agricultural Research; Guy Vergères, PhD Dr, Principal Investigator — Agroscope Liebefeld-Posieux Research Station ALP; Marjukka Kolehmainen, Principal Investigator — University of Eastern Finland; Sandra Wallner, Principal Investigator — Med Uni Graz; Cristina Andres-Lacueva, Principal Investigator — University of Barcelona
Locations (12):
- Medizinische Universität Graz, Graz, Austria
- University of Leuven (KU Leuven), Leuven, Belgium
- Charles University Prague, Prague, Czechia
- University of Copenhagen, Copenhagen, Denmark
- University of Eastern Finland, Kuopio, Finland
- INRA - L'Institut Nationel de la Recherche Agronomique, Clermont, France
- University College Dublin, Dublin, Ireland
- CRA-NUT - Centro di Ricerca per gli Alimenti e la Nutrizione, Rome, Italy
- TNO, Zeist, Gelderland, Netherlands
- University of Barcelona, Barcelona, Spain
- Agroscope, Institute for Food Sciences, Bern, Switzerland
- Newcastle University, Newcastle, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
An internal review board, consisting of Principal Investigators from all participating countries, will review all data requests.
  A data request format is available that should be used for filing such a request. The format requires stating the research questions that should be answered with the requested data, type of data, populations requirements (exclusion criteria), data analysis and public disclosure.
  All study participants have the ability to withdraw their data from use for answering specific research questions at any time.